CLINICAL TRIAL: NCT05081180
Title: Single-arm, Multicenter Phase I/Ib Study of Avelumab + Lenvatinib in Children With Primary CNS Tumors
Brief Title: Study of Avelumab in Combination With Lenvatinib for Children With Primary CNS Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS100070_0087; 2020-004397-22 (EudraCT Number); 2024-512940-51-00 (Other: EU CTIS)
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Central Nervous System Tumors
Keywords: Avelumab; Lenvatinib; Tumors; Pediatric CNS tumors
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasms | interventions — avelumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab + Lenvatinib (Experimental)
  Interventions: Drug: Avelumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Avelumab — Participants with primary CNS malignancies who have received at least 1 prior therapy will be enrolled into Dose Escalation Part 1 and will receive intravenous infusion at a flat dose or weight based dose of Avelumab, every 2 weeks (Q2W) until progression, unacceptable toxicity, or withdrawal of consent. Enrollment into part 1 of the study will end when Maximum tolerated dose (MTD) and/or a safe Recommended Dose for Expansion (RDE) for the expansion cohort is determined. Participants with defined CNS tumors will be enrolled into Dose Expansion Part 2 and will receive RDE in Part 2 until progression, unacceptable toxicity, or withdrawal of consent.
Drug: Lenvatinib — Participants with primary CNS malignancies who have received at least 1 prior therapy will be enrolled into Dose Escalation Part 1 and will receive daily oral escalated dose level of Lenvatinib until progression, unacceptable toxicity, or withdrawal of consent. Enrollment into part 1 of the study will end when MTD and/or a safe Recommended Dose for Expansion (RDE) for the expansion cohort is determined. Participants with defined CNS tumors will be enrolled into Dose Expansion Part 2 and will receive RDE of Lenvatinib in Part 2 until progression, unacceptable toxicity, or withdrawal of consent.

SUMMARY:
This study consists of 2 parts: Dose Escalation Part 1 and Dose Expansion Part 2. The Dose Escalation Part 1 will evaluate the safety and tolerability of Avelumab in combination with Lenvatinib and determine the recommended Avelumab and Lenvatinib dose for expansion. Dose Expansion Part 2 will assess the efficacy of Avelumab in combination with Lenvatinib by Progression-free Survival in participants with pre-defined primary central nervous system (CNS) tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed diagnosis of primary CNS malignancy as follows: a) Primary CNS tumors: the tumor should be considered high-grade histologically; prior radiotherapy is allowed; participants must have progressed after at least 1 prior systemic therapy, except for those with diffuse midline glioma with or without the H3 K27M mutation. b) Specific for participants with diffuse midline glioma with or without the H3 K27M mutation: prior radiotherapy is allowed; no more than 1 prior systemic therapy is allowed; participants with diffuse midline glioma with or without the H3 K27M mutation who have not received prior systemic therapy but have prior radiotherapy only are allowed to enroll
* On screening scans, measurable disease by RANO criteria
* Participants must have a Lansky performance status >= 50 for age <= 16 years or Karnofsky performance status >= 50 for age > 16 years at Screening
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with low-grade gliomas, for example but not limited to, subependymal giant cell astrocytoma, pilocytic astrocytoma and World Health organization (WHO) Grade 1 tumors
* Participants demonstrating evidence of worsening of neurologic deficit within 1 week prior to initiation of study interventions
* Participants with bulky tumor, defined as: a) Tumor with any evidence of uncal herniation or midline shift; b) Tumor with a diameter of > 4 centimeters (cm) in 1 dimension on T2/ fluid-attenuated inversion recovery (FLAIR) images; c) Tumor that in the opinion of the Investigator shows significant mass effect
* Participants are not eligible if they experience uncontrolled seizures, defined as: a) Seizures requiring regular use of rescue medications. b) Seizures requiring increasing doses of antiepileptic medications. c) Seizures that in the opinion of the Investigator compromise the ability of the participant to tolerate study intervention or interfere with study procedures
* Participants who have received major surgery (including but not limited to neurosurgical resection, brain biopsy, or radiation to the primary brain tumor) within 28 days prior to the first dose of study interventions
* Participants with history of intracranial hemorrhage/spinal cord hemorrhage within 28 days prior to the first dose of study interventions
* Other protocol defined exclusion criteria could apply

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Part 1: Number of Participants with Common Terminology Criteria for Adverse Events (CTCAE) Grade Greater Than or Equal to (>=) 3 Treatment-emergent Adverse Event (TEAEs) According to National Cancer Institute-CTCAE Version 5.0 | up to 857 days
Dose Escalation Part 1: Number of Participants With Dose Limiting Toxicities (DLTs) | Baseline (Day 1) up to Day 28
Dose Expansion Part 2: Progression-free Survival (PFS) According to Response Assessment in Neuro-Oncology (RANO) Criteria as Assessed by Investigators | until progressive disease or death, assessed up to Day 1534

SECONDARY OUTCOMES:
Dose Escalation Part 1: Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Treatment-related Adverse Events (AEs), Adverse Event of Special Interest (AESIs), AEs Leading to Deaths | up to 876 days
Dose Escalation Part 1: Number of Participants with Treatment-Emergent Adverse Events (AEs) Based on Severity According to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | up to 876 days
Dose Escalation Part 1: Number of Participants with Clinically Significant Changes from Baseline in Laboratory Parameters | up to 876 days
Dose Escalation Part 1: Objective Response Rate (ORR) According to Response Assessment in Neuro-Oncology (RANO) Criteria as Assessed by Investigators | up to 876 days
Dose Escalation Part 1: Duration of Response (DOR) According to Response Assessment in Neuro-Oncology (RANO) Criteria as Assessed by Investigators | up to 876 days
Dose Escalation Part 1: Progression-Free Survival (PFS) According to Response Assessment in Neuro-Oncology (RANO) Criteria | until progressive disease or death, assessed up to 876 days
Dose Escalation Part 1: Overall Survival (OS) | up to 876 days
Dose Escalation Part 1: Serum Observed Concentration at End of Infusion (CEOI) of Avelumab | Pre-dose up to 30 days after last dose, assessed up to approximately 876 days
Dose Escalation Part 1: Area Under the Serum Concentration-Time Curve From the Time of Dosing 336 Hours (AUC0-336 [hr]) of Avelumab | Pre-dose up to 336 hours post-dose, assessed up to approximately 876 days
Dose Escalation Part 1: Serum Concentration Observed Immediately Before Next Dosing (Ctrough) of Avelumab | Pre-dose up to 30 days after last dose, assessed up to approximately 876 days
Dose Escalation Part 1: Maximum Observed Plasma Concentration (Cmax) of Lenvatinib | Pre-dose up to 30 days after last dose, assessed up to approximately 876 days
Dose Escalation Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Lenvatinib | Pre-dose up to 30 days after last dose, assessed up to approximately 876 days
Dose Escalation (Part 1): Area Under the Plasma Concentration-Time Curve From the Time of Dosing to 24 Hours (AUC0-24 [hr]) of Lenvatinib: | Pre-dose up to 24 hours post-dose, assessed up to approximately 876 days
Dose Escalation Part 1: Immunogenicity of Avelumab as Measured by Antidrug Antibody (ADA) Assay | up to 876 days
Dose Expansion Part 2: Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Treatment-related Adverse Events (AEs), Adverse Event of Special Interest (AESIs), AEs Leading to Deaths | up to Day 1534
Dose Expansion Part 2: Number of Participants with Treatment-Emergent Adverse Events (AEs) Based on Severity According to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | up to Day 1534
Dose Expansion Part 2: Number of Participants with Clinically Significant Changes in Laboratory Parameters | up to Day 1534
Dose Expansion Part 2: Objective Response Rate (ORR) Rate According to Response Assessment in Neuro-Oncology (RANO) Criteria as Assessed by Investigators | up to Day 1534
Dose Expansion Part 2: Duration of Response (DOR) According to Response Assessment in Neuro-Oncology (RANO) Criteria as Assessed by Investigators | up to Day 1534
Dose Expansion Part 2: Overall Survival (OS) | up to Day 1534
Dose Expansion Part 2: Serum Observed Concentration at End of Infusion (CEOI) of Avelumab | Pre-dose up to 30 days after last dose, assessed up to approximately Day 1534
Dose Expansion Part 2:Serum Concentration Observed Immediately Before Next Dosing (Ctrough) of Avelumab | Pre-dose up to 30 days after last dose, assessed up to approximately Day 1534
Dose Expansion Part 2: Maximum Observed Plasma Concentration (Cmax) of Lenvatinib | Pre-dose up to 30 days after last dose, assessed up to approximately Day 1534
Dose Expansion Part 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Lenvatinib | Pre-dose up to 30 days after last dose, assessed up to approximately Day 1534
Dose Expansion Part 2: Immunogenicity of avelumab as measured by ADA assay | up to Day 1534

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (9):
- Canada (2):
  - CHU Sainte-Justine, Montreal
  - The Hospital for Sick Children, Toronto
- France (3):
  - CHU Angers - Hôpital Hôtel Dieu - Service de Cancérologie Pédiatrique, Angers
  - Hôpital de la Timone, Marseille
  - Institut Curie - Centre de Lutte Contre le Cancer (CLCC) de Paris, Paris
- Germany (2):
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Muenster, Münster
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS100070_0087
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html